CLINICAL TRIAL: NCT04979091
Title: Low Testosterone and High Estradiol Are Associated With Disease Severity in Critically Ill COVID-19 Patients - a Retrospective Analysis
Brief Title: Sex Hormone Dysregulations Are Associated With Critical Illness in COVID-19 Patients
Acronym: HAM-SEX-C19
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government)
Responsible Party: Sponsor
Other Study IDs: HAM-SEX-C19
Record Dates: First submitted 2021-07-25; First posted 2021-07-27 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Critical Illness
Keywords: ICU, COVID-19, testosteron, estradiol, sex-hormone
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sex Hormones — A panel of 13 hormones was measured in plasma samples of COVID-19 patients (total testosterone, free testosterone, dihydrotestosterone, androstenedione, 17-β-estradiol, estrone, sex hormone-binding globulin, thyroid-stimulating hormone, free triiodothyronine (T3), free thyroxine (T4), luteinizing hormone, follicle-stimulating hormone and cortisol).

SUMMARY:
Males develop more severe SARS-CoV-2 infection related disease outcome than females. Herein, sex hormones were repeatedly proposed to play an important role in Covid-19 pathophysiology and immunity. However, it is yet unclear whether sex hormones are associated with Covid-19 outcome in males and females. In this study, we analyzed sex hormones, cytokine and chemokine responses as well as performed a large profile analysis of 600 metabolites in critically-ill male and female Covid-19 patients in comparison to healthy controls and patients with coronary heart diseases as a prime Covid-19 comorbidity. We here show that dysregulated sex hormones, IFN-γ levels and unique metabolic signatures are associated with critical illness in Covid-19 patients. Both, male and female Covid-19 patients, present elevated estradiol levels which positively correlates with IFN-γ levels.

Male Covid-19 patients additionally display severe testosterone and triglyceride deficiencies as compared to female patients and healthy controls. Our results suggest that male Covid-19 patients suffer from multiple metabolic disorders, which may lead to higher risk for fatal outcome. These findings will help to understand molecular pathways involved in Covid-19 pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Admission on ICU
* Covid-19

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill Covid-19 patients and Critically ill Non-Covid-19 patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-08 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Sex hormone in critical ill COVID-19 patients | Day at admission
  testosterone
Sex hormone in critical ill COVID-19 patients | Day at admission
  estradiol
Sex hormone in critical ill COVID-19 patients | Day at admission
  sex hormone-binding globulin
Sex hormone in critical ill patients | Day at admission
  testosterone
Sex hormone in critical ill patients | Day at admission
  estradiol

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, Prof., Study Chair — University Medical Center Hamburg-Eppendorf, Germany
Locations (1):
- University Medical Center, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Preprint — https://www.medrxiv.org/content/10.1101/2020.05.07.20073817v2